CLINICAL TRIAL: NCT00973219
Title: A Randomized Prospective Open-label Trial for Comparing Combination Therapy Peg-Interferon Alfa-2a/Adefovir Dipivoxil and Peg-Interferon Alfa-2a/Tenofovir Disoproxil Fumarate Versus no Treatment in HBeAg Negative Chronic Hepatitis B Patients With Low Viral Load.
Brief Title: Hepatitis B Surface Antigen(HBsAg) Loss in Chronic Hepatitis B Patients With Low Viral Load
Acronym: LVL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, H.W.Reesink, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTM16002; EudraCT number: 2009-013117-94; ABR number: 28338
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Chronic Hepatitis B
Keywords: HBsAg loss; HBsAg seroconversion; chronic hepatitis B; low viral load; inactive carrier hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Peg-Interferon alfa 2a + Adefovir (Active Comparator): 50 HBeAg negative chronic hepatitis B patients with low viral load will receive Peg-Interferon alfa 2a + Adefovir for a period of 48 weeks.
  Interventions: Drug: Peg-Interferon alfa 2a + Adefovir dipivoxil, Peg-Interferon alfa 2a + Tenofovir disoproxil fumarate
- Peg-Interferon alfa 2a + Tenofovir (Active Comparator): 50 HBeAg negative chronic hepatitis B patients with low viral load will receive Peg-Interferon alfa 2a + Tenofovir for a period of 48 weeks.
  Interventions: Drug: Peg-Interferon alfa 2a + Adefovir dipivoxil, Peg-Interferon alfa 2a + Tenofovir disoproxil fumarate
- no treatment (No Intervention): 50 HBeAg negative chronic hepatitis B patients with low viral load will not receive treatment during a period of 48 weeks

INTERVENTIONS:
Drug: Peg-Interferon alfa 2a + Adefovir dipivoxil, Peg-Interferon alfa 2a + Tenofovir disoproxil fumarate — Peg-Interferon alfa 2a 180ug/week + Adefovir dipivoxil 10mg/day, Peg-Interferon alfa 2a 180ug/week + Tenofovir disoproxil fumarate 245mg/day
  Other Names: Pegsys®; Hepsera®; Viread®
  Arms: Peg-Interferon alfa 2a + Adefovir; Peg-Interferon alfa 2a + Tenofovir

SUMMARY:
Rationale:

Worldwide, approximately 400 million people are chronically infected with hepatitis B virus (HBV). Chronic HBV infection increases the risk of developing cirrhosis, hepatic decompensation and hepatocellular carcinoma (HCC). The risk of developing hepatocellular carcinoma is highest in HBeAg positive patients with high HBV DNA levels, but still the relative risk remains 10 for HBeAg negative patients. Furthermore it has been shown that when HBsAg is cleared before cirrhosis has developed, the prognosis is excellent. Recently the investigators have shown that HBeAg negative patients with high HBV-DNA load and low baseline HBsAg levels had a significantly higher HBsAg clearance (positive predictive value of 85%) after combination therapy with peginterferon alfa2a (Peg-IFN) and adefovir.

Based on these results, a trial was designed to investigate whether combination of a nucleos(t)ide analogue combined with PegIFN, could also provoke a high rate of HBsAg clearance in chronic hepatitis B patients with low (HBV DNA <20,000 IU/mL) viral load.

Study design:

This is a three arm open-label prospective randomized controlled trial. 150 patients will be enrolled into the study after assessment of eligibility. All patients must have documented HBsAg positivity for longer than 6 months, HBeAg negativity, anti-HBe positivity, HBV DNA < 20,000 IU/mL and ALT < 5 * upper limit of normal. Patients with a Child Pugh class B or C will be excluded. Group 1 will consist of patients treated with Peg-IFN and adefovir, group 2 will consist of patients treated with Peg-IFN and tenofovir and group 3 will consist of untreated controls. Patients in group 1 and 2 will receive medication for the period of one year. For enrolment into the study a liverbiopsy at time of enrolment is compulsory and is advisable at end of treatment (week 48).

Study population: The study population will consist of 150 patients chronically infected with hepatitis B virus with low viral load and HBeAg negativity.

Main study parameters/endpoints:

The aim of this study is to investigate what proportion of HBeAg negative, inactive carriers of the hepatitis B virus with low (< 20,000 IU/mL) load will lose HBsAg when treated with nucleot(s)ide analogue/Peg-IFN combination therapy.

In this study the investigators hypothesize that both treatment with peg-interferon and ADF or Peg-IFN and TDF in HBeAg negative chronic hepatitis B patients with low HBV DNA viral load will induce a high rate of HBsAg loss, comparable to that in patients with high viral load after treatment with ADF and Peg-IFN.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients > 18 and ≤ 70 years of age
* Positive HBsAg for more than 6 months.
* Negative for HBeAg for more than 6 months.
* HBV DNA < 2.0 E04 IU/mL
* Serum ALT < 5 * ULN as determined by two values taken >14 days apart during the six months before the first dose of study drug with at least one of the determinations obtained during the screening period.
* Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug.

Exclusion Criteria:

* Patients co-infected with HCV, HIV or who have decompensated liver disease, hepato-cellular carcinoma, significant cardiac disease, significant renal disease, seizure disorders or severe retinopathy.
* Patients who have received nucleos(t)ide analogues for their chronic hepatitis B within 6 weeks before enrollment or have received Peg-IFN within 3 months before enrollment.
* Patients must not have received any other systemic anti-viral, anti-neoplastic or immuno-modulatory treatment (including supraphysiologic doses of steroids or radiation) <3 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* Positive test at screening for anti-HAV IgM, anti-HIV, HCV RNA. (Patients that have cleared the hepatitis C virus can be included in the study)
* Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation in the study are also excluded. Exception: patients who have had a limited (<7 day) course of acyclovir for herpetic lesions more than 1 month prior to the first administration of test drug are not excluded.
* Evidence of decompensated liver disease (Child pugh B-C)
* Serum total bilirubin > twice the upper limit of normal at screening
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease.
* History or other evidence of a medical condition associated with chronic liver disease other than HBV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver diseases including Wilson's disease and alfa1-antitrypsin deficiency, alcoholic liver disease, toxin exposures, thalassemia).
* Women with ongoing pregnancy or who are breast feeding.
* Neutrophil count <1500 cells/mm3 or platelet count <80,000 cells/mm3 at screening.
* Hemoglobin < 7.1 mmol/L (< 11.5 g/dL) for females and < 7.8 mmol/L (< 12.5 g/dL) for men at screening.
* Serum creatinine level >1.5 times the upper limit of normal at screening.
* Unstable ongoing severe psychiatric disease, especially depression (stable patients can be included).
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis).
* History or other evidence of chronic pulmonary and cardiac disease associated with functional limitation. Severe cardiac disease (e.g., NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases).
* History of a severe seizure disorder or current anticonvulsant use and clinically unstable disease.
* Evidence of an active or suspected cancer or a history of malignancy where the risk of recurrence is >20% within 5 years. Patients with a lesion suspicious of hepatic malignancy on a screening imaging study will only be eligible if the likelihood of carcinoma is <10% following an appropriate evaluation.
* Major organ transplantation. (patients with skin, cornea or bone transplantation are allowed to be included into the study)
* Thyroid disease with thyroid function poorly controlled on prescribed medications. Patients with elevated thyroid stimulating hormone or T4 concentrations, with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease that are not stable on prescribed medication are excluded. Stable patients can be included.
* History or other evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration) or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
* Patients with a value of alfa-fetoprotein >100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months.
* Evidence of current hard drug(s) (i.e. cannabis products are allowed) and/or alcohol abuse (20g/day for women and 30g/day for men).
* Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is to demonstrate the efficacy of combination therapy (Peg-IFN and adefovir or Peg-IFN and tenofovir) for inducing loss of HBsAg compared to no-treatment in HBeAg negative chronic hepatitis B patients with low viral load. | 6.5 years including long term follow up

SECONDARY OUTCOMES:
The secondary objectives are to evaluate: a. the rate of HBsAg loss and anti-HBs seroconversion, b. To establish predictive markers at baseline and during the first 12 weeks of treatment for response of primary and secondary endpoints. | 6.5 years including long term follow up.

CONTACTS AND LOCATIONS:
Overall Officials: H.R. Reesink, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] de Niet A, Jansen L, Stelma F, Willemse SB, Kuiken SD, Weijer S, van Nieuwkerk CMJ, Zaaijer HL, Molenkamp R, Takkenberg RB, Koot M, Verheij J, Beuers U, Reesink HW. Peg-interferon plus nucleotide analogue treatment versus no treatment in patients with chronic hepatitis B with a low viral load: a randomised controlled, open-label trial. Lancet Gastroenterol Hepatol. 2017 Aug;2(8):576-584. doi: 10.1016/S2468-1253(17)30083-3. Epub 2017 May 15. PMID 28522204